CLINICAL TRIAL: NCT04118335
Title: The Effect of Oral Care by Black Mulberry Syrup on Oral Mucositis in Individuals With COPD
Brief Title: Mulberry Syrup on Oral Mucositis Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/42
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Oral Mucositis
Keywords: Oral mucositis in COPD patients; complementary therapies; nursing interventions; oral care with black mulberry syrup
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The individuals in the intervention group were asked to gargle with 5 ml black mulberry syrup three times a day after meals and wait average one minute in the mouth and then swallow, in addition to the standard practice of the clinic. According to the standard practice of the clinic, mucositis treatment was performed by nystatin and/or benzidamine hydrochloride to the patients with the request of the physician. The patients were followed for 15 days. The 15-day period is consistent with the duration of mucositis healing in the literature. Follow-up and evaluation of patients who were discharged early were performed by home visits and made a phone call everyday.
  Interventions: Other: Black Mulberry Syrup
- Control Group (No Intervention): Standard procedures of the clinic were applied to control group. According to the standard practice of the clinic, mucositis treatment was performed by nystatin and/or benzidamine hydrochloride to the patients with the request of the physician. Follow-up and evaluation of patients who were discharged early were performed by home visits and made a phone call everyday.

INTERVENTIONS:
Other: Black Mulberry Syrup — The individuals in the intervention group gargled with 5 ml black mulberry syrup and waited average one minute and then swallow it.
  Arms: Intervention Group

SUMMARY:
Objective: This study was carried out to investigate the effectiveness of oral care with black mulberry syrup on oral mucositis healing in individuals with COPD.

Study Design: The quantitative part of the study was conducted as a randomized controlled experimental study, the qualitative section was conducted by in-depth interview method. The study was performed with 40 patients who were hospitalized in the Chest Diseases Clinic. In addition to the standard practice of the clinic, the individuals in the intervention group gargled with 5 ml black mulberry syrup and waited average one minute and then swallow it. They did this application 3 times a day after meals. 10 individuals in the intervention group were interviewed by using a semi-structured interview form.

DETAILED DESCRIPTION:
Objective: This mix study was carried out to investigate the effectiveness of oral care with black mulberry syrup on oral mucositis healing in individuals with COPD.

Study Design: The quantitative part of the study was conducted as a randomized controlled experimental study, the qualitative section was conducted by in-depth interview method. Approval from the Ethics Committee and written permission from the institution were obtained. After the participants were informed about the purpose of the study, their written consents were obtained. The study was performed with 40 patients who were hospitalized in the Chest Diseases Clinic. In addition to the standard practice of the clinic, the individuals in the intervention group gargled with 5 ml black mulberry syrup and waited average one minute and then swallow it. They did this application 3 times a day after meals. 10 individuals in the intervention group were interviewed by using a semi-structured interview form.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* no visual or hearing problem,
* unimpaired time and place orientation,
* no psychiatric disorders,
* diagnosed with COPD,
* oral mucositis developed,
* used Nystatin and/or Benzidamine Hydrochloride therapy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Duration of oral mucositis healing | Change from oral mucositis healing levels at 15 days
  Oral mucosa of patients were evaluated with The Oral Evaluation Guide by examining the patients mucous membrane with the help of light source and asking patients.
  Oral Evaluation Guide: The guideline evaluates the changes of the oral mucosa in eight areas. In the evaluation of the guide, numerical expressions like 1, 2, 3 are used and the changes in voice, swallowing function, saliva, tongue, lips, mucous membranes, gums, teeth or prostheses are scored. When scoring, all scores from eight areas are collected and the Oral Mucosal Score (OMS) is calculated. The lowest possible score is 8 and the highest score is 24. As the score increases, intra-oral complaints and the severity of mucositis increase.

SECONDARY OUTCOMES:
Severity of oral mucositis | Change from severity of oral mucositis at 15 days
  Severity of oral mucositis were evaluated with World Health Organization Oral Mucositis Scoring Index by examining the patients mucous membrane with the help of light source and asking patients.
  World Health Organization Oral Mucositis Scoring Index: According to this index, the severity of oral mucositis is graded as grade 0; no mucositis, grade 1; mild, grade 2; moderate, grade 3-4; severe mucositis.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Korkut, PhD, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No